CLINICAL TRIAL: NCT03675477
Title: A Phase II Randomized, Placebo Controlled, Double-blind, 4 Arms Dose-ranging Study to Evaluate the Efficacy and Safety of SHR0302 Compared to Placebo in Patients With Moderate to Severe Active Ulcerative Colitis.
Brief Title: A Phase II Study in Patients With Moderate to Severe Active Ulcerative Colitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSJ10101; 2018-003364-31 (EudraCT Number)
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SHR0302 8mg QD (Experimental): Participants randomized in this arm will receive SHR0302 8mg QD for the treatment phase. All participants that had completed the 8-week treatment phase (non-responders or responders) had the option to enter a blinded 8-week extension phase to continue to receive SHR0302 8mg QD.
  Those who had completed the first 8-week of the treatment phase, but decided not to enter into the extension phase were also required to attend the 2-week follow-up visit. Participants who immaturely withdrew during the first treatment phase could not enter the extension phase.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
  Interventions: Drug: SHR0302
- SHR0302 4mg BD (Experimental): Participants randomized in this arm will receive SHR0302 4mg BD for the treatment phase. All participants that had completed the 8-week treatment phase (non-responders or responders) had the option to enter a blinded 8-week extension phase to continue to receive SHR0302 4mg BD.
  Those who had completed the first 8-week of the treatment phase, but decided not to enter into the extension phase were also required to attend the 2-week follow-up visit. Participants who immaturely withdrew during the first treatment phase could not enter the extension phase.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
  Interventions: Drug: SHR0302
- SHR0302 4mg QD (Experimental): Participants randomized in this arm will receive SHR0302 4mg QD for the treatment phase. All participants that had completed the 8-week treatment phase (non-responders or responders) had the option to enter a blinded 8-week extension phase to continue to receive SHR0302 4mg QD.
  Those who had completed the first 8-week of the treatment phase, but decided not to enter into the extension phase were also required to attend the 2-week follow-up visit. Participants who immaturely withdrew during the first treatment phase could not enter the extension phase.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
  Interventions: Drug: SHR0302
- placebo (Placebo Comparator): Participants randomized in this arm will receive the placebo until week 8, and then will be re-randomized into one of the 3 active arms ( 4mg QD, 4mg BD, 8mg QD of SHR0302) in a 1:1:1 allocation ratio until the end of the study at week 16.
  Those who had completed the first 8-week of the treatment phase, but decided not to enter into the extension phase were also required to attend the 2-week follow-up visit. Participants who immaturely withdrew during the first treatment phase could not enter the extension phase.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
  Placebos: Placebo Oral Tablet
  Interventions: Drug: SHR0302; Drug: Placebo

INTERVENTIONS:
Drug: SHR0302 — The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a Janus kinase inhibitor).
  Other Names: Ivarmacitinib
Drug: Placebo — Placebo Oral Tablet
  Arms: placebo

SUMMARY:
The proposed study is a randomized, double-blind,placebo-controlled, multicenter phase II study to investigate the safety and efficacy of SHR0302 in patients with moderate to severe active ulcerative colitis. The study aims to evaluate the optimal dose of SHR0302 and time needed to induce clinical response in active ulcerative colitis patients.

This is an 8+8 weeks study, in which participants who complete the first 8 weeks treatment phase, will have the option to enter a blinded active arms 8-week extension phase. Early withdrawn subjects during the first treatment phase can not enter the extension phase. The total duration of the study participation, including extension and follow-up, will be approximately 18 weeks.

SHR0302 is a Janus kinase 1(JAK1) inhibitor, capable of blocking Janus kinase-signal transducer and activator of transcription (JAK-STATs) pathway and controlling inflammation. Therefore it has the potential to be a treatment for ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subject age ≥ 18 and ≤75 years of age at randomization.
* Active ulcerative colitis with a 9-point modified Mayo score of 5 to 9 points and endoscopic subscore of 2 to 3 (The duration of the time between endoscopy and baseline should not exceed 10 days and allow central over read turn over before randomization).
* Subject should have at least three-month history of Ulcerative Colitis diagnosis at randomization.

Exclusion Criteria:

* Diagnosis of indeterminate colitis, or clinical findings suggestive of Crohn's disease.
* Subjects with ulcerative colitis, which is confined to a proctitis (distal 15 cm or less).
* Treatment naïve subjects diagnosed with ulcerative colitis (without previous exposure to treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, Study Director — Reistone Pharma
Locations (66):
- United States (3):
  - Wellness Clinical Research, LLLC-Central Florida, Lake Wales, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Tampa, Florida
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
- China (35):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Baotou Central Hospital, Baotou, Inner Mongalia
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Peking University Shougang Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jillin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Fujian Provincial Hospital, Fuzhou
  - The Sixth Affiliated Hospital of Sun Yat- Sen University, Guangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Huaian First People's Hospital, Huai'an
  - Huzhou Central Hospital, Huzhou
  - Qilu Hospital of Shandong University, Jinan
  - The First People's Hospital of Lianyungang, Lianyungang
  - Jiangsu Province Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Pingxiang People's Hospital, Pingxiang
  - Shanghai East Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
  - Shanxi Provincial People's Hospital, Taiyuan
  - Second Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Union Medical Center, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital Affiliated to Tongji Medicine College, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Yijishan Hospital of Wannan Medical College, Wuhu
- Poland (12):
  - Indywidualma Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Amicare Sp. z o.o. Sp.k, Lodz
  - IP Clinic, Lodz
  - NZOZ Almedica, Nowy Targ
  - SOLUMED Centrum Medyczne, Poznan
  - KO-MED Centra Kliniczne Plulawy, Puławy
  - Specjalistyczna Praktyka Lekarska dr med. Marek Horynski, Sopot
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Nzoz Formed, Wadowice
  - Nzoz Vivamed, Warsaw
  - PlanetMed sp. z o.o., Wroclaw
- Wellness Clinical Research, LLC, Vega Baja, Puerto Rico
- Ukraine (15):
  - RCI Chernivtsi Regional Clinical Hospital Dept of Gastroenterology Bukovinsky SMU, Chernivtsi
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Central City Clinical Hospital Dept of Theraphy No. 2 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - Ivana -Frankivsk Hospital, Ivano-Frankivsk
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - CI Karabelesh Kherson CCH, Kherson
  - Kherson City Clinical Hospital, Kherson
  - Khmelnytska Regional Hospital, Khmelnytskyi
  - Kyiv City Clinical Hospital #1, Kyiv
  - Kyiv Railway Clinical Hospital #2 of Branch "Health Center" of the Public Joint Stock Company "Ukrai, Kyiv
  - CNE of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv
  - Vinnytsia M.I.Pyrogov Regional Clinical Hospital, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - CI City Clinical Hospital #6 Dept of Gastroenterology, Zaporizhzhia
  - O.F. Herbachevskiyi Zhytomyr Regional Clinical Hospital, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen B, Zhong J, Li X, Pan F, Ding Y, Zhang Y, Chen H, Liu F, Zhang Z, Zhang L, Drozda R, Oliinyk O, Goh AH, Chen X, Sun X, Rubin DT, Sandborn WJ, Chen M. Efficacy and Safety of Ivarmacitinib in Patients With Moderate-to-Severe, Active, Ulcerative Colitis: A Phase II Study. Gastroenterology. 2022 Dec;163(6):1555-1568. doi: 10.1053/j.gastro.2022.08.007. Epub 2022 Aug 10. PMID 35963369

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Started | 41 | 41 | 41 | 41
Completed | 41 | 41 | 41 | 41
Not Completed | 0 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Started | 47 (11 participants in the placebo arm in the treatment phase were randomized into the 8mg QD arm in the extension phase. 36 participants in the 8mg QD arm in the treatment phase remained in the same dose group in the extension phase.) | 49 (10 participants in the placebo arm in the treatment phase were randomized into the 4mg BD arm in the extension phase. 39 participants in the 4mg BD arm in the treatment phase remained in the same dose group in the extension phase.) | 48 (13 participants in the placebo arm in the treatment phase were randomized into the 4mg QD arm in the extension phase. 35 participants in the 4mg QD arm in the treatment phase remained in the same dose group in the extension phase.) | 0
Completed | 47 | 49 | 48 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo | Total
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (13.3) | 40.3 (12.3) | 39.6 (10.0) | 42.7 (12.9) | 40.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 13 | 22 | 64
  Male | 27 | 26 | 28 | 19 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 29 | 25 | 25 | 24 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 16 | 16 | 17 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Time since initial primary diagnosis [Mean (Standard Deviation); unit: years] | 5.05 (4.16) | 5.62 (5.62) | 5.17 (5.17) | 5.77 (5.19) | 5.40 (5.03)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subject Achieve Clinical Response at Week 8
Description: Clinical response is defined as a decrease from baseline in a 9-point modified Mayo score of at least 2 points and at least 30%, with an accompanying reduction in the subscore for rectal bleeding of at least 1 point or absolute subscore for rectal bleeding of 0 or 1.
  The 9-point modified Mayo score is the Mayo score excluding the Physician Global Assessment sub-score, hence the maximum is 9 points and the minimum is 0 point, includes:
  Stool Frequency 0 = Normal
  1. = 1-2 stools/day more than normal
  2. = 3-4 stools/day more than normal
  3. = 5 or more stools/day than normal
  Rectal bleeding 0 = None
  1. = Visible blood with stool less than half the time
  2. = Visible blood with stool half of the time or more
  3. = Passing blood alone
  Mucosal appearance at endoscopy 0 = Normal or inactive disease
  1. = Mild disease (erythema, decreased vascular pattern, mild friability
  2. = Moderate disease (marked erythema, absent vascular pattern, friability, erosio
Time Frame: Week 8
Measure: Number; unit: percentage of participants
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Number analyzed (Participants) | 41 | 41 | 41 | 41
percentage of participants | 46.3 | 46.3 | 43.9 | 26.8

2. Secondary Outcome: The Percentage of Subjects Achieve Clinical Remission
Description: Clinical remission was defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point. The percentage of subjects who achieve clinical remission per 9-point modified Mayo score at week 8, where stool frequency subscore ≤ 1, rectal bleeding subscore of 0, and endoscopic subscore ≤ 1.
  9-point modified Mayo score includes: Stool Frequency 0 = Normal
  1. = 1-2 stools/day more than normal
  2. = 3-4 stools/day more than normal
  3. = 5 or more stools/day than normal
  Rectal bleeding 0 = None
  1. = Visible blood with stool less than half the time
  2. = Visible blood with stool half of the time or more
  3. = Passing blood alone
  Mucosal appearance at endoscopy 0 = Normal or inactive disease
  1. = Mild disease (erythema, decreased vascular pattern, mild friability
  2. = Moderate disease (marked erythema, absent vascular pattern, friability, erosions)
  3. = Severe disease (spontaneous bleeding, ulceration)
Time Frame: Week 8
Measure: Number; unit: percentage of participants
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Number analyzed (Participants) | 41 | 41 | 41 | 41
percentage of participants | 22.0 | 24.4 | 24.4 | 4.9

3. Secondary Outcome: The Percentage of Subjects Achieve Clinical Remission at Week 8
Description: Clinical remission was defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point. The percentage of subjects achieve clinical remission at week 8 as per a total Mayo score of 2 points or lower ≤2, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0.
  The 9-point modified Mayo score includes:
  Stool Frequency 0 = Normal
  1. = 1-2 stools/day more than normal
  2. = 3-4 stools/day more than normal
  3. = 5 or more stools/day than normal
  Rectal bleeding 0 = None
  1. = Visible blood with stool less than half the time
  2. = Visible blood with stool half of the time or more
  3. = Passing blood alone
  Mucosal appearance at endoscopy 0 = Normal or inactive disease
  1. = Mild disease (erythema, decreased vascular pattern, mild friability
  2. = Moderate disease (marked erythema, absent vascular patt
Time Frame: Week 8
Measure: Number; unit: percentage of participants
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Number analyzed (Participants) | 41 | 41 | 41 | 41
percentage of participants | 14.6 | 17.1 | 17.1 | 2.4

4. Secondary Outcome: The Percentage of Subjects Achieve Endoscopic Remission (Mucosal Healing) at Week 8
Description: Endoscopic remission was defined by Mayo endoscopic subscore ≤ 1 point. Mayo endoscopic subscore defines score 0 as normal or inactive disease, score 1 as mild disease (erythema, decreased vascular pattern, mild friability); score 2 as moderate disease (marked erythema, absent vascular pattern, friability, erosions)； score 3 as severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 8
Measure: Number; unit: percentage of participants
Arm/Group | SHR0302 8mg QD | SHR0302 4mg BD | SHR0302 4mg QD | Placebo
Number analyzed (Participants) | 41 | 41 | 41 | 41
percentage of participants | 26.8 | 29.3 | 36.6 | 14.6

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: All participants that had completed the 8-week treatment phase (non-responders or responders) had the option to enter a blinded 8-week extension phase to receive the active drug. In the extension phase, participants randomized into placebo in the treatment phase were randomized into one of the three active groups above (4mg QD, 4mg BD, and 8mg QD) in a 1:1:1 ratio. Participants randomized to the active arms in the treatment phase remained in the same dose group in the extension phase.
Groups:
- Treatment Phase-SHR0302 8mg QD: Participants randomized in this arm will receive dose A of SHR0302 until the end of the study at week 16.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
- Treatment Phase-SHR0302 4mg BD: Participants randomized in this arm will receive dose B of SHR0302 until the end of the study at week 16.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
- Treatment Phase-SHR0302 4mg QD: Participants randomized in this arm will receive dose C of SHR0302 until the end of the study at week 16.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
- Treatment Phase-Placebo: Participants randomized in this arm will receive placebo of SHR0302 until the end of the study at week 16.
  SHR0302: The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK (known as a JAK inhibitor).
- Extension Phase-SHR0302 8mg QD → SHR0302 8mg QD; Extension Phase-SHR0302 4mg BD → SHR0302 4mg BD; Extension Phase-SHR0302 4mg QD → SHR0302 4mg QD; Extension Phase-placebo → SHR0302 8mg QD; Extension Phase-placebo → SHR0302 4mg BD; Extension Phase-placebo → SHR0302 4mg QD: All participants that had completed the 8-week treatment phase (non-responders or responders) had the option to enter a blinded 8-week extension phase to receive active drug. In the extension phase, participants randomized into placebo in the treatment phase were randomized into one of the three active groups above (dose A, dose B, and dose C) in a 1:1:1 ratio. Participants randomized to the active arms in the treatment phase remained in the same dose group in the extension phase.
Arm/Group | Treatment Phase-SHR0302 8mg QD | Treatment Phase-SHR0302 4mg BD | Treatment Phase-SHR0302 4mg QD | Treatment Phase-Placebo | Extension Phase-SHR0302 8mg QD → SHR0302 8mg QD | Extension Phase-SHR0302 4mg BD → SHR0302 4mg BD | Extension Phase-SHR0302 4mg QD → SHR0302 4mg QD | Extension Phase-placebo → SHR0302 8mg QD | Extension Phase-placebo → SHR0302 4mg BD | Extension Phase-placebo → SHR0302 4mg QD
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/41 | 0/36 | 0/39 | 0/35 | 0/11 | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/41 | 0/41 | 2/41 | 2/41 | 1/36 | 0/39 | 0/35 | 1/11 | 1/10 | 0/13
Other Adverse Events (participants affected / at risk) | 13/41 | 11/41 | 12/41 | 7/41 | 13/36 | 8/39 | 11/35 | 5/11 | 5/10 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase-SHR0302 8mg QD (N=41) | Treatment Phase-SHR0302 4mg BD (N=41) | Treatment Phase-SHR0302 4mg QD (N=41) | Treatment Phase-Placebo (N=41) | Extension Phase-SHR0302 8mg QD → SHR0302 8mg QD (N=36) | Extension Phase-SHR0302 4mg BD → SHR0302 4mg BD (N=39) | Extension Phase-SHR0302 4mg QD → SHR0302 4mg QD (N=35) | Extension Phase-placebo → SHR0302 8mg QD (N=11) | Extension Phase-placebo → SHR0302 4mg BD (N=10) | Extension Phase-placebo → SHR0302 4mg QD (N=13)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase-SHR0302 8mg QD (N=41) | Treatment Phase-SHR0302 4mg BD (N=41) | Treatment Phase-SHR0302 4mg QD (N=41) | Treatment Phase-Placebo (N=41) | Extension Phase-SHR0302 8mg QD → SHR0302 8mg QD (N=36) | Extension Phase-SHR0302 4mg BD → SHR0302 4mg BD (N=39) | Extension Phase-SHR0302 4mg QD → SHR0302 4mg QD (N=35) | Extension Phase-placebo → SHR0302 8mg QD (N=11) | Extension Phase-placebo → SHR0302 4mg BD (N=10) | Extension Phase-placebo → SHR0302 4mg QD (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 3 | 2 | 0 | 2 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03675477/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03675477/SAP_001.pdf